CLINICAL TRIAL: NCT02647164
Title: The Value Of Circulating Tumor Cells In Patient With NSCLC In Postoperative Recurrence Monitoring
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: GenoSaber (Industry)
Responsible Party: Sponsor
Other Study IDs: CTC2015-01
Record Dates: First submitted 2015-12-28; First posted 2016-01-06 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2015-09

CONDITIONS: Non-small-cell Lung Carcinoma
Keywords: Non-small-cell lung carcinoma; Circulating tumor cells
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to assess the value of circulating tumor cells (CTC)for non-small cell lung cancer in the postoperative recurrence monitoring by comparing the CTCs, CT and tumor markers at different time points.The time of CTC and carcinoembryonic antigen(CEA) detection is baseline, 2~7 days, 3 months, 6 months, 12 months, 24 months, 36 months after the surgery. And the time of CT detection is 6 months, 12 months, 24 months, 36 months after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years old
* Patients with histologically documented (stage Ⅰ/Ⅱ/ⅢA ) non-small cell lung cancer.
* Patients will undergo surgery.
* Patients with preoperative CTCs ≥8.5 Units / 3 ml
* Informed consent must be obtained from all patients prior to beginning therapy. Patients should have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients with histologically documented not (stage Ⅰ/Ⅱ/ⅢA ) non-small cell lung cancer.
* After the operation review, patients' result of CTC, CT and tumor markers is incomplete at the same point.
* The blood sample isn't collected in predetermined time.
* The blood samples appear hemolysis.
* The blood sample isn't enough.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with NSCLC(stage Ⅰ/Ⅱ/ⅢA), who will receive operation.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Circulating tumor cells will be detected by Immunomagnetic negative screening and targeted PCR method. | 3 years

SECONDARY OUTCOMES:
carcinoembryonic antigen(CEA) concentration will be detected by electrochemical luminescence. | 3 years
Liconography using conventional CT examination results. | 3 years